CLINICAL TRIAL: NCT01412307
Title: A Phase 1/2 Study of Lenalidomide in Combination With Bendamustine (LEBEN) in Relapsed and Primary Refractory Hodgkin Lymphoma
Brief Title: A Phase 1/2 Study of Lenalidomide in Combination With Bendamustine in Relapsed and Primary Refractory Hodgkin Lymphoma
Acronym: LEBEN
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Principal Investigator, Antonio Pinto, Director of Hematology Oncology and Stem Cell Transplant Unit at National Tumor Institute 'Fondazione G. Pascale', Naples - Italy, Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale
Organization: GiovanniPascale (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEBEN-HL; 2011-002810-35 (EudraCT Number)
Record Dates: First submitted 2011-08-03; First posted 2011-08-09 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Recurrent Adult Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; Lenalidomide; Bendamustine; Salvage therapy; Palliation
MeSH Terms: conditions — Hodgkin Disease | interventions — Lenalidomide; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide plus bendamustine (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Bendamustine; Other: Bio-specimen Retention

INTERVENTIONS:
Drug: Lenalidomide — 10, 15, 20 or 25 mg orally per cohort day 1-28 in a 28 days cycle
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: Bendamustine — intravenous on days 1, 8 and 15 of each 28-days cycle at fixed dose of 60 mg/m2, as a 30-60 min i.v. infusion
  Other Names: SDX-105; Ribomustin; Treanda; Cytostasan
Other: Bio-specimen Retention — Samples with DNA and without DNA

SUMMARY:
Management of patients with recurring Hodgkin lymphoma (HL) after stem cell transplantation failure represents a typical unmet medical need prompting active development and validation of new agents and treatment strategies. The LEBEN protocol combines two agents, lenalidomide and bendamustine, framing different targets on both tumor and microenvironmental cells of HL. These agents, while showing a low risk of overlapping extrahematologic toxicities, may hit the proliferation machinery of H-RS cells and/or their progenitors, synergistically inhibit tumor-related angiogenesis and interfere on cytokine-mediate circuitries operating in the microenvironment to support tumor cell survival.

A weekly schedule of bendamustine, at 60 mg/m2, is combined with the continuous administration of increasing dose of lenalidomide (10, 15, 20 e 25 mg dose levels in a 28-day cycle). Such schedule of Bendamustine is aimed at enhancing the antiangiogenic and immunomodulatory activity of continuous Lenalidomide, as studies have shown that low and protracted doses of alkylators induce a decrease in microvascular density of tumor tissues and inhibit mobilization and viability of circulating endothelial progenitors.

The Bayesian phase 1/2 dose finding method of Thall and Cook was employed. This method chooses doses based-on both response and toxicity, and accounts for the trade-off between these two outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed classical Hodgkin lymphoma (HL).
* Patients must have failed an autologous stem cell transplant or be ineligible for high-dose therapy due to chemorefractory disease (as defined as <50% response to standard salvage chemotherapy), age or comorbidity.
* Patients must have at least one target PET-avid bidimensionally measurable lesion,
* Age >18 years
* Life expectancy of greater than 3 months
* ECOG performance status <2
* Patients must have adequate organ and marrow function as defined below: absolute neutrophil count >1,000/mL; platelets >75,000/mL; total bilirubin < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's disease); however dose reduction is recommended for Bendamustine in patients with 30 - 70 % tumour involvement of the liver and moderately diminished liver function (serum bilirubin 1.2 - 3.0 mg/dl); AST(SGOT)/ALT(SGPT) <3 X institutional upper limit of normal; creatinine within normal institutional limits OR creatinine clearance >50 mL/min/1.73 m2
* Patients must have echocardiogram or gated blood pool scan (MUGA) with an ejection fraction > or = to 50%
* If patients have a history of malignancy other than cutaneous basal cell or squamous cell carcinoma, they must be disease-free for ~ 5 years at the time of enrolment
* Patients must accept contraception measures until 4 weeks after the completion of chemotherapy, and up to 6 months for male patients.
* Women of child-bearing must have a medically supervised negative pregnancy test even if had been using effective contraception.
* Patients agree not to share study medication with another person and to return all unused study drug to the investigator
* Patients or their guardians must be capable to understand and must be willing to sign a written informed consent document.

Exclusion Criteria:

* Treatment with chemotherapy or external radiotherapy within 6 weeks, or monoclonal antibodies within 8 weeks or radioimmunoconjugates in the previous 12 weeks prior to entering the study
* Treatment with any other investigational agent
* Parenchymal brain or leptomeningeal HL involvement
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used in the study
* Known HIV positivity or active infectious hepatitis, type A, B, or C
* Clinically significant cardiac disease (NYHA Class III or IV)
* Abnormal QTcF interval prolonged (> 459 msec)
* Known pregnancy or breastfeeding.
* Jaundice
* Yellow fever vaccination
* Medical illness unrelated to HL, which in the opinion of the attending physician and principal investigator will preclude safe administration of lenalidomide and bendamustine
* Corticoid treatment different from low dose prednisone or methylprednisone (up to 16 mg), used for B symptoms control.
* Contraindications for receiving prophylaxis against deep vein thrombosis
* Thromboembolic disease grade 3-4 in the last 6 months
* More than one month between staging procedures and the start of the treatment
* Major surgical procedures less than 30 days before the start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Dose finding, as best trade-off between toxicity and efficacy according to the Bayesian phase I/II dose finding method of Thall and Cook | Evaluation at day +56, i.g. after two cycles.
  According to the Bayesian phase I/II dose finding method of Thall and Cook,a target efficacy-toxicity trade-off contour has been constructed by fitting a curve to target values of pE (probability ofEfficacy) and pT (probability of Toxicity) of 0.30 and 0.40, respectively and probability cut-offs pE (for Efficacy)and pT (for Toxicity) set at 0.10 and 0.10,respectively.The area underneath the target contour has desirable πE, πT pairs. Up to 36 patients can be treated in cohorts of size 3. The 'best' dose is defined as that giving the largest response-toxicity trade-off.

SECONDARY OUTCOMES:
AE/SAE rate at completion of treatment | After course 6. i.g. about 6 months
Overall Rate Response | After 2, 4 and 6 cycles
Event Free Survival | From the time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason
Time to Progression | From entry until documented lymphoma progression or death as a result of lymphoma.
Response Duration | From the time when criteria for response (i.g. CR or PR) are met, for which the event is the first documentation of relapse or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pinto, MD, Principal Investigator — Hematology Oncology and Stem Cell Transplantation Unit , IRCCS Fondazione "G.Pascale" - Naples, Italy; Gaetano Corazzelli, MD, Principal Investigator — Hematology Oncology and Stem Cell Transplantation Unit , IRCCS Fondazione "G.Pascale" - Naples, Italy
Locations (1):
- Hematology Oncology and Stem Cell Transplantation Unit , IRCCS Fondazione "G.Pascale", Naples, Italy

REFERENCES:
- [Result] http://meetinglibrary.asco.org/content/132091-144